CLINICAL TRIAL: NCT01783444
Title: A Three-arm, Randomized, Open Label, Phase II Study of Everolimus in Combination With Exemestane Versus Everolimus Alone Versus Capecitabine in the Treatment of Postmenopausal Women With Estrogen Receptor Positive, Locally Advanced, Recurrent, or Metastatic Breast Cancer After Recurrence or Progression on Prior Letrozole or Anastrozole.
Brief Title: A Phase II Study of Everolimus in Combination With Exemestane Versus Everolimus Alone Versus Capecitabine in Advance Breast Cancer.
Acronym: BOLERO-6
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRAD001Y2201; 2012-003757-28 (EudraCT Number)
Record Dates: First submitted 2013-01-11; First posted 2013-02-05 (Estimated); Results first posted 2021-02-26 (Actual); Last update posted 2021-02-26 (Actual); Status verified 2021-02

CONDITIONS: Breast Cancer
Keywords: Everolimus; Exemestane; Capecitabine; locally advanced; metastatic; breast cancer; breast cancer positive for human epidermal growth factor receptor 2; HER2; HER2 positive; breast cancer progression; estrogen-receptor positive breast cancer; ER
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis | interventions — Capecitabine; exemestane; Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Capecitabine 1250 mg/m2 (Experimental): Capecitabine (1250 mg/m2 twice daily) for two weeks, followed by one week rest period in 3-weeks cycles (investigational arm).
  Interventions: Drug: Capecitabine
- Everolimus 10 mg (Experimental): Everolimus (10 mg daily) (investigational arm).
  Interventions: Drug: Everolimus
- Everolimus 10 mg + Exemestane 25 mg (Active Comparator): Everolimus (10 mg daily) with Exemestane (25 mg daily) (control arm).
  Interventions: Drug: Exemestane; Drug: Everolimus

INTERVENTIONS:
Drug: Capecitabine — Capecitabine, tablets for oral use, 1250 mg/m² twice daily for 2 weeks followed by one week rest (3-week-cycle) (locally supplied)
  Other Names: Capecitabine monotherapy
  Arms: Capecitabine 1250 mg/m2
Drug: Exemestane — Exemestane, tablets for oral use, 25 mg per day in (locally supplied)
  Other Names: Control arm
  Arms: Everolimus 10 mg + Exemestane 25 mg
Drug: Everolimus — Everolimus, 5 mg tablets for oral use, 10 mg (2 x 5 mg) per day (centrally supplied)
  Other Names: Everolimus monotherapy; RAD001
  Arms: Everolimus 10 mg; Everolimus 10 mg + Exemestane 25 mg

SUMMARY:
This was a three-arm, randomized, open label, multi-center phase II study investigating the combination of everolimus (10mg daily) with exemestane (25mg daily) versus everolimus (10mg daily) versus capecitabine (1250mg/m2 twice daily for 14 days, 3-week cycle) in patients with estrogen-receptor positive, HER2 negative, advanced breast cancer after recurrence or progression on letrozole or anastrozole.

DETAILED DESCRIPTION:
The reference therapy (control arm) used in the course of this trial was the combination arm of everolimus plus exemestane. The investigational therapies in the context of this study were everolimus monotherapy and capecitabine monotherapy. All treatments were taken orally until disease progression, intolerable toxicity or withdrawal of patient's informed consent. Patients were randomly assigned with equal allocation to one of the treatment arms:

1. Exemestane (25mg daily) in combination with everolimus (10mg daily)
2. Everolimus (10mg daily)
3. Capecitabine (1250mg/m2 twice daily) orally for two weeks, followed by a one week rest period in 3-weeks cycles.

Treatment assignment was stratified by the presence of visceral disease (yes vs. no). Visceral refered to lung, liver, heart, ovary, spleen, kidney, adrenal gland, malignant pleural or pericardial effusion or malignant ascites.

Randomization and Treatment Phase:

At Visit 3 all eligible patients were randomized in 1:1:1 ratio to receive everolimus (10mg daily oral tablets) in combination with exemestane (25 mg daily oral tablets), everolimus (10mg daily oral tablets) or capecitabine monotherapy (1250mg/m2 twice daily orally for two weeks followed by a one week rest period in 3-weeks cycles). Assignment was stratified by the presence of visceral disease (yes vs. no). Visceral refered to lung, liver, heart, ovary, spleen, kidney, adrenal gland, malignant pleural or pericardial effusion or malignant ascites. After randomization, study treatment started and continued until progression, intolerable toxicity or consent withdrawal. Further treatment after progression and study treatment discontinuation was at the investigator's discretion. Dose adjustment (reduction, interruption) according to safety findings was allowed. Regular safety and efficacy reviews by Data Monitoring Committee (DMC) were performed. Tumor assessments were performed every 6 weeks until disease progression. Additional evaluation were performed to confirm response at 4 weeks after it was first observed. After at least 150 PFS events had been documented per RECIST 1.1 by local assessment in each of the two following groups: (i) everolimus + exemestane arm plus everolimus monotherapy arm, and (ii) everolimus + exemestane arm plus capecitabine monotherapy arm, the frequency of tumor assessments was changed to every 12 weeks or as clinically indicated.

Follow-up phase:

Patients were followed for safety for 30 days after study treatment discontinuation. If a patient did not discontinue study treatment due to disease progression, lost to follow-up or consent withdrawal, then tumor assessments continued to be performed every 6 weeks until disease progression, death, lost to follow-up or investigator decision in patient best interest.

Survival Data Collection:

All patients were followed for survival status at least every 3 months regardless of treatment discontinuation reason and up to two years after randomization of last patient. Survival information could be obtained via phone and information were documented in the source documents and eCRF. Additional survival follow-up might be performed more frequently if a survival update was required for reporting the results or to meet safety or regulatory needs.

ELIGIBILITY:
Key Inclusion Criteria:

- Women with locally advanced, recurrent, or metastatic breast cancer along with confirmation of estrogen-receptor positive (ER+). Measurable disease defined as at least one lesion ≥ 10 mm by CT or MRI that can be accurately measured in at least one dimension (CT scan slice thickness ≤ 5 mm) OR • Bone lesions: lytic or mixed (lytic + blastic) in the absence of measurable disease as defined above.

Key Exclusion Criteria:

- Patients who received more than one chemotherapy line. Patients with only non-measurable lesions other than lytic or mixed (lytic and blastic) bone metastasis.Previous treatment with exemestane, mTOR inhibitors, PI3K inhibitors or AKT inhibitors.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 309 (Actual)
Dates: Start 2013-02-26 (Actual); Primary Completion 2018-07-02 (Actual); Study Completion 2018-07-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (81):
- United States (19):
  - University of California at Los Angeles Mattel Children's Hospital, Los Angeles, California
  - Sharp Memorial Hospital SharpClinicalOncologyResearch, San Diego, California
  - Florida Cancer Specialists Dept of Oncology (2), Fort Myers, Florida
  - Florida Cancer Specialists FL Cancer Specialists, Fort Myers, Florida
  - Lahey Clinic Dept of Lahey Clinic (2), Burlington, Massachusetts
  - New England Hematology/ Oncology Associates, P.C. SC, Newton, Massachusetts
  - Glacier View Research Institute - Cancer SC, Kalispell, Montana
  - Trinitas Comprehensive Cancer Center SC, Elizabeth, New Jersey
  - Hackensack University Medical Center Dept of Oncology, Hackensack, New Jersey
  - Rutgers-New Jersey Medical School SC, Newark, New Jersey
  - Oncology Hematology Care Inc Oncology Hematology Care 2, Cincinnati, Ohio
  - Oklahoma Cancer Specialists and Research Institute Oklahoma Cancer Specialists, Tulsa, Oklahoma
  - Chattanooga Oncology and Hematology Assoicates, PC Chattanooga Oncology, Chattanooga, Tennessee
  - The Jones Clinic SC, Germantown, Tennessee
  - University of Tennessee SC, Knoxville, Tennessee
  - Sarah Cannon Research Institute SC (2), Nashville, Tennessee
  - The Center for Cancer and Blood Disorders Dept. of The Ctr for C & BD, Fort Worth, Texas
  - University of Virginia Health Systems SC-4, Charlottesville, Virginia
  - Northwest Medical Specialties Dept of Onc, Tacoma, Washington
- Argentina (5):
  - Novartis Investigative Site, CABA, Buenos Aires
  - Novartis Investigative Site, Posadas, Misiones Province
  - Novartis Investigative Site, Rosario, Santa Fe Province
  - Novartis Investigative Site, Rio Negro, Viedma
  - Novartis Investigative Site, Córdoba
- Australia (4):
  - Novartis Investigative Site, Randwick, New South Wales
  - Novartis Investigative Site, Wahroonga, New South Wales
  - Novartis Investigative Site, Malvern, Victoria
  - Novartis Investigative Site, Parkville, Victoria
- Novartis Investigative Site, Liège, Belgium
- Brazil (5):
  - Novartis Investigative Site, Salvador, Estado de Bahia
  - Novartis Investigative Site, Natal, Rio Grande do Norte
  - Novartis Investigative Site, Passo Fundo, Rio Grande do Sul
  - Novartis Investigative Site, Porto Alegre, Rio Grande do Sul
  - Novartis Investigative Site, São Paulo, São Paulo
- Denmark (6):
  - Novartis Investigative Site, Aarhus
  - Novartis Investigative Site, Copenhagen
  - Novartis Investigative Site, Næstved
  - Novartis Investigative Site, Odense C
  - Novartis Investigative Site, Roskilde
  - Novartis Investigative Site, Vejle
- Hungary (3):
  - Novartis Investigative Site, Budapest, HUN
  - Novartis Investigative Site, Debrecen
  - Novartis Investigative Site, Tatabánya
- India (4):
  - Novartis Investigative Site, Hyderabad, Andhra Pradesh
  - Novartis Investigative Site, Pune, Maharashtra
  - Novartis Investigative Site, Kolkata, West Bengal
  - Novartis Investigative Site, Mumbai
- Ireland (3):
  - Novartis Investigative Site, Limerick, Co Limerick
  - Novartis Investigative Site, Dublin
  - Novartis Investigative Site, Galway
- Lebanon (4):
  - Novartis Investigative Site, Beirut
  - Novartis Investigative Site, El Achrafiyé
  - Novartis Investigative Site, Hazmiyeh
  - Novartis Investigative Site, Saida
- Malaysia (2):
  - Novartis Investigative Site, Kota Kinabalu, Sabah
  - Novartis Investigative Site, Kuala Lumpur
- Peru (4):
  - Novartis Investigative Site, Jesus Maria, Lima region
  - Novartis Investigative Site, San Borja, Lima region
  - Novartis Investigative Site, Surquillo, Lima region
  - Novartis Investigative Site, Arequipa
- Russia (3):
  - Novartis Investigative Site, Arkhangelsk
  - Novartis Investigative Site, Moscow
  - Novartis Investigative Site, Saint Petersburg
- Spain (3):
  - Novartis Investigative Site, Seville, Andalusia
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, Madrid
- Sweden (6):
  - Novartis Investigative Site, Eskilstuna
  - Novartis Investigative Site, Jönköping
  - Novartis Investigative Site, Stockholm
  - Novartis Investigative Site, Uppsala
  - Novartis Investigative Site, Vaxjo
  - Novartis Investigative Site, Västerås
- Thailand (3):
  - Novartis Investigative Site, Lopburi, Changwat Lop Buri
  - Novartis Investigative Site, Songkhla, Hat Yai
  - Novartis Investigative Site, Muang
- Turkey (Türkiye) (3):
  - Novartis Investigative Site, Adana
  - Novartis Investigative Site, Istanbul
  - Novartis Investigative Site, Izmir
- United Kingdom (3):
  - Novartis Investigative Site, East Kilbride
  - Novartis Investigative Site, Middlesbrough
  - Novartis Investigative Site, Nottingham

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com
URL: https://www.clinicalstudydatarequest.com/

REFERENCES:
- [Derived] Jerusalem G, de Boer RH, Hurvitz S, Yardley DA, Kovalenko E, Ejlertsen B, Blau S, Ozguroglu M, Landherr L, Ewertz M, Taran T, Fan J, Noel-Baron F, Louveau AL, Burris H. Everolimus Plus Exemestane vs Everolimus or Capecitabine Monotherapy for Estrogen Receptor-Positive, HER2-Negative Advanced Breast Cancer: The BOLERO-6 Randomized Clinical Trial. JAMA Oncol. 2018 Oct 1;4(10):1367-1374. doi: 10.1001/jamaoncol.2018.2262. PMID 29862411

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 84 centers in 18 countries worldwide: Belgium (1), Denmark (6), Hungary (3), Ireland (3), Spain (4), Sweden (6), United Kingdom (3), United States (19), Argentina (6), Brazil (5), Peru (4), India (4), Lebanon (5), Malaysia (2), Russia (3), Thailand (3), Turkey (3) Australia (4)
Pre-assignment Details: A total of 300 subjects were planned and total of 309 subjects were randomized to everolimus plus exemestane (control arm) (N = 104), everolimus alone (N = 103), or capecitabine (N = 102).
Period: Treatment Phase
Arm/Group | Everolimus 10 mg + Exemestane 25 mg | Everolimus 10 mg | Capecitabine 1250 mg/m2
Started (All randomized subjects (FAS)) | 104 | 103 | 102
Safety Set (At least 1 dose of study treatment and a 1 post baseline safety assessment) | 104 | 103 | 102
Completed | 0 | 0 | 0
Not Completed | 104 | 103 | 102
Not completed — Adverse Event | 9 | 20 | 19
Not completed — Disease Progression | 76 | 66 | 64
Not completed — Death | 2 | 2 | 2
Not completed — Protocol Violation | 1 | 1 | 2
Not completed — Withdrawal by Subject | 6 | 8 | 9
Not completed — Administrative problems | 2 | 0 | 1
Not completed — Physician Decision | 8 | 6 | 5
Period: Post-Treatment Efficacy Follow-Up Phase
Arm/Group | Everolimus 10 mg + Exemestane 25 mg | Everolimus 10 mg | Capecitabine 1250 mg/m2
Started (All patients who discontinued treatment and entered Post-Treatment Efficacy Follow-Up Phase) | 96 (All patients who entered Post-Treatment Efficacy Follow-Up Phase) | 93 (All patients who entered Post-Treatment Efficacy Follow-Up Phase) | 91 (All patients who entered Post-Treatment Efficacy Follow-Up Phase)
Completed | 0 | 0 | 0
Not Completed | 96 | 93 | 91
Not completed — Disease Progression | 7 | 8 | 11
Not completed — Death | 9 | 7 | 5
Not completed — Withdrawal by Subject | 4 | 8 | 8
Not completed — Administrative Problems | 0 | 1 | 0
Not completed — New cancer therapy | 7 | 16 | 15
Not completed — Followup phase completed as per protocol | 69 | 53 | 52

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Everolimus 10 mg + Exemestane 25 mg | Everolimus 10 mg | Capecitabine 1250 mg/m2 | Total
Number analyzed (Participants) | 104 | 103 | 102 | 309
Age, Continuous [Mean (Standard Deviation); unit: Years] | 60.9 (10.47) | 61.3 (9.08) | 59.7 (10.50) | 60.6 (10.03)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 104 | 103 | 102 | 309
  Male | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: Participants]
  Caucasian | 78 | 85 | 91 | 254
  Black | 1 | 2 | 0 | 3
  Asian | 11 | 8 | 8 | 27
  Native American | 3 | 2 | 0 | 5
  Other | 11 | 6 | 3 | 20
ECOG Performance Status [Count of Participants; unit: Participants]
  No Restrictions | 54 | 48 | 57 | 159
  Only Light Work | 42 | 50 | 39 | 131
  Only Self Care | 5 | 3 | 4 | 12
  Missing | 3 | 2 | 2 | 7

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS) - Everolimus Plus Exemestane Versus Everolimus Alone
Description: Progression Free Survival (PFS) is defined as the time from date of randomization to the date of first radiologically documented progression or death due to any cause. If a patient did not have an event, PFS was censored at the date of the last adequate tumor assessment. PFS was compared between the everolimus + exemestane combination therapy with the everolimus monotherapy.
Time Frame: Date of randomization to the date of first documented tumor progression or death from any cause, whichever occurs first, reported between day of first patient randomized up to 39 months
Population: Full Analysis Set (FAS), which consisted of all randomized patients, was considered.
Measure: Median (90% Confidence Interval); unit: Months
Arm/Group | Everolimus 10 mg + Exemestane 25 mg | Everolimus 10 mg
Number analyzed (Participants) | 104 | 103
Months | 8.41 [6.60 to 9.72] | 6.77 [5.52 to 7.20]
Statistical Analysis 1: Comparison: Everolimus 10 mg + Exemestane 25 mg vs Everolimus 10 mg; Test type: Non-Inferiority — Hazard ratio obtained from stratified Cox model (stratified by presence/absence of visceral metastasis as per IWRS); Hazard Ratio (HR) = 0.74, 90% CI 2-sided [0.57 to 0.97]

2. Secondary Outcome: Progression Free Survival (PFS) - Everolimus Plus Exemestane Versus Capecitabine Alone
Description: as for outcome 1
Time Frame: as for outcome 1
Population: Full Analysis Set (FAS), which consisted of all randomized patients, was considered.
Measure: Median (90% Confidence Interval); unit: Months
Arm/Group | Everolimus 10 mg + Exemestane 25 mg | Capecitabine 1250 mg/m2
Number analyzed (Participants) | 104 | 102
Months | 8.41 [6.60 to 9.72] | 9.59 [8.25 to 15.05]
Statistical Analysis 1: Comparison: Everolimus 10 mg + Exemestane 25 mg vs Capecitabine 1250 mg/m2; Test type: Non-Inferiority — Hazard ratio obtained from stratified Cox model (stratified by presence/absence of visceral metastasis as per IWRS); Hazard Ratio (HR) = 1.26, 90% CI 2-sided [0.96 to 1.66]

3. Secondary Outcome: Overall Survival (OS)
Description: Overall Survival (OS) is defined as the time from date of randomization to date of death due to any cause. If a patient was not known to have died by the date of analysis cut-off, OS was censored at the date of last known date patient alive.
Time Frame: Every 3 months following end of treatment visit, assessed for approximately 54 months
Population: Full Analysis Set (FAS), which consisted of all randomized patients, was considered.
Measure: Median (90% Confidence Interval); unit: Months
Arm/Group | Everolimus 10 mg + Exemestane 25 mg | Everolimus 10 mg | Capecitabine 1250 mg/m2
Number analyzed (Participants) | 104 | 103 | 102
Months | 23.06 [19.48 to 27.96] | 29.27 [24.28 to 31.77] | 25.56 [23.82 to 33.35]
Statistical Analysis 1: Comparison: Everolimus 10 mg + Exemestane 25 mg vs Everolimus 10 mg; Test type: Non-Inferiority — Hazard ratio obtained from stratified Cox model (stratified by presence/absence of visceral metastasis as per IWRS); Hazard Ratio (HR) = 1.27, 90% CI 2-sided [0.95 to 1.70]
Statistical Analysis 2: Comparison: Everolimus 10 mg + Exemestane 25 mg vs Capecitabine 1250 mg/m2; Test type: Non-Inferiority — Hazard ratio obtained from stratified Cox model (stratified by presence/absence of visceral metastasis as per IWRS); Hazard Ratio (HR) = 1.33, 90% CI 2-sided [0.99 to 1.79]

4. Secondary Outcome: Overall Response Rate (ORR)
Description: Overall Response Rate (ORR) as the proportion of patients whose best overall response is either complete response (CR) or partial response (PR) according to RECIST 1.1 This was assessed in the full patient population. Complete response is achieved when all lesions evaluated at baseline are absent at subsequent visit. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR. Only descriptive statistics.
Time Frame: From the date of randomization until the date of the first documented disease progression or date of death from any cause whichever came first, assessed for approximately 43 months
Population: Full Analysis Set (FAS), which consisted of all randomized patients, was considered.
Measure: Number (90% Confidence Interval); unit: Percentage of Participants
Arm/Group | Everolimus 10 mg + Exemestane 25 mg | Everolimus 10 mg | Capecitabine 1250 mg/m2
Number analyzed (Participants) | 104 | 103 | 102
Percentage of Participants | 21 [13.9 to 27.8] | 12 [6.9 to 18.2] | 23 [15.9 to 30.4]

5. Secondary Outcome: Clinical Benefit Rate (CBR)
Description: Clinical Benefit Rate (CBR) is defined as the proportion of participants with a best overall response of complete response (CR) or partial response (PR) or stable disease (SD) or Non-CR/non-PD lasting more than 24 weeks based on local investigator's assessment according to RECIST 1.1. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR, Stable disease (SD), neither sufficient shrinkage to qualify for PR or CR nor an increase in lesions which would qualify for PD; CBR = CR+PR+SD. Only descriptive statistics.
Time Frame: as for outcome 4
Population: Full Analysis Set (FAS), which consisted of all randomized patients, was considered.
Measure: Number (90% Confidence Interval); unit: Percentage of Participants
Arm/Group | Everolimus 10 mg + Exemestane 25 mg | Everolimus 10 mg | Capecitabine 1250 mg/m2
Number analyzed (Participants) | 104 | 103 | 102
Percentage of Participants | 59 [48.2 to 65.0] | 43 [33.5 to 50.3] | 53 [43.4 to 60.5]

6. Secondary Outcome: Time to Eastern Cooperative Oncology Group (ECOG) Performance Deterioration
Description: The Eastern Cooperative Oncology Group (ECOG) Performance Status is a scale used to assess physical health of subjects,ranging from 0 (most active) to 5 (least active). Definitive deterioration is defined as no improvement in the ECOG status following observation of the deterioration.
Time Frame: Baseline, every 6 weeks up to about 43 months
Population: Full Analysis Set (FAS), which consisted of all randomized patients, was considered.
Measure: Median (90% Confidence Interval); unit: Weeks
Arm/Group | Everolimus 10 mg + Exemestane 25 mg | Everolimus 10 mg | Capecitabine 1250 mg/m2
Number analyzed (Participants) | 104 | 103 | 102
Weeks | 72.57 [38.71 to NA] — NA: Not estimable due to high number of censors primarily due to treatment discontinuation. | 126.57 [72.14 to NA] — NA: Not estimable due to high number of censors primarily due to treatment discontinuation | 120.00 [72.57 to NA] — NA: Not estimable due to high number of censors primarily due to treatment discontinuation
Statistical Analysis 1: Comparison: Everolimus 10 mg + Exemestane 25 mg vs Everolimus 10 mg; Test type: Non-Inferiority — Hazard ratio obtained from stratified Cox model (stratified by presence/absence of visceral metastasis as per IWRS); Hazard Ratio (HR) = 1.09, 90% CI 2-sided [0.72 to 1.66]
Statistical Analysis 2: Comparison: Everolimus 10 mg + Exemestane 25 mg vs Capecitabine 1250 mg/m2; Test type: Non-Inferiority — Hazard ratio obtained from stratified Cox model (stratified by presence/absence of visceral metastasis as per IWRS); Hazard Ratio (HR) = 1.18, 90% CI 2-sided [0.78 to 1.77]

7. Secondary Outcome: Time to 10% Definitive Deterioration in the Global Health Status / Quality of Life
Description: The global health status/QoL scale score of the QLQ-C30 is identified as the primary PRO variable of interest. Physical Functioning (PF), Emotional Functioning (EF) and Social Functioning (SF) scale scores of the QLQ-C30. The time to definitive 10% deterioration is the number of days between the date of randomization and the date of the assessment at which definitive deterioration is seen. Definitive 10% (5-point) deterioration is defined as a decrease in score by at least 10% (5-points) compared to baseline, with no later increase above this threshold observed during the course of the study.
Time Frame: Baseline, every 6 weeks up to about 43 months
Population: Full Analysis Set (FAS), which consisted of all randomized patients, was considered.
Measure: Median (90% Confidence Interval); unit: Weeks
Arm/Group | Everolimus 10 mg + Exemestane 25 mg | Everolimus 10 mg | Capecitabine 1250 mg/m2
Number analyzed (Participants) | 104 | 103 | 102
Weeks | 30.86 [24.29 to 78.00] | 23.86 [12.57 to 24.71] | 61.29 [36.86 to 143.71]
Statistical Analysis 1: Comparison: Everolimus 10 mg + Exemestane 25 mg vs Everolimus 10 mg; Test type: Non-Inferiority — Hazard ratio obtained from stratified Cox model (stratified by presence/absence of visceral metastasis as per IWRS); Hazard Ratio (HR) = 0.64, 90% CI 2-sided [0.46 to 0.88]
Statistical Analysis 2: Comparison: Everolimus 10 mg + Exemestane 25 mg vs Capecitabine 1250 mg/m2; Test type: Non-Inferiority — Hazard ratio obtained from stratified Cox model (stratified by presence/absence of visceral metastasis as per IWRS); Hazard Ratio (HR) = 1.33, 90% CI 2-sided [0.93 to 1.91]

8. Secondary Outcome: Mean Change in Treatment Satisfaction Questionnaire for Medication (TSQM) Between Week 3 and 12
Description: TSQM was used to measure the Patients' self-reported satisfaction or dissatisfaction with the study treatment. The differences in mean scale scores between weeks 3 and 12 comparing treatment satisfaction in the different treatment arms: everolimus + exemestane combination therapy versus everolimus monotherapy, and everolimus + exemestane combination therapy versus capecitabine monotherapy. The TSQM version 1.4 domain scores range from 0 to 100 with higher scores representing a higher satisfaction on that domain.
Time Frame: Week 3, Week 12
Population: Full Analysis Set (FAS), which consisted of all randomized patients, was considered. Only participants who had both post-baseline assessments were included.
Measure: Mean (Standard Deviation); unit: Unit on a scale
Arm/Group | Everolimus 10 mg + Exemestane 25 mg | Everolimus 10 mg | Capecitabine 1250 mg/m2
Number analyzed (Participants) | 104 | 103 | 102
Unit on a scale
  Side-effects: number analyzed (Participants) | 68 | 59 | 59
  Side-effects | -4.8 (28.88) | -9.1 (21.88) | -2.6 (22.45)
  Effectiveness: number analyzed (Participants) | 63 | 58 | 57
  Effectiveness | -2.2 (20.15) | 1.2 (26.51) | 1.2 (21.61)
  Convenience: number analyzed (Participants) | 68 | 60 | 56
  Convenience | -0.6 (12.00) | 1.0 (16.41) | 0.5 (17.67)
  Global satisfaction: number analyzed (Participants) | 66 | 60 | 56
  Global satisfaction | -1.0 (17.32) | 1.8 (20.80) | 2.3 (16.96)
Statistical Analysis 1: Comparison: Everolimus 10 mg + Exemestane 25 mg vs Everolimus 10 mg; Side-effects; Test type: Other; Mean Difference (Net) = 4.3, 90% CI 2-sided [-3.3 to 11.9]
Statistical Analysis 2: Comparison: Everolimus 10 mg + Exemestane 25 mg vs Capecitabine 1250 mg/m2; Side-effects; Test type: Other; Mean Difference (Net) = -2.2, 90% CI 2-sided [-9.9 to 5.5]
Statistical Analysis 3: Comparison: Everolimus 10 mg + Exemestane 25 mg vs Everolimus 10 mg; Effectiveness; Test type: Other; Mean Difference (Net) = -3.3, 90% CI 2-sided [-10.4 to 3.8]
Statistical Analysis 4: Comparison: Everolimus 10 mg + Exemestane 25 mg vs Capecitabine 1250 mg/m2; Effectiveness; Test type: Other; Mean Difference (Net) = -3.3, 90% CI 2-sided [-9.7 to 3.0]
Statistical Analysis 5: Comparison: Everolimus 10 mg + Exemestane 25 mg vs Everolimus 10 mg; Convenience; Test type: Other; Mean Difference (Net) = -1.6, 90% CI 2-sided [-5.8 to 2.5]
Statistical Analysis 6: Comparison: Everolimus 10 mg + Exemestane 25 mg vs Capecitabine 1250 mg/m2; Convenience; Test type: Other; Mean Difference (Net) = -1.1, 90% CI 2-sided [-5.5 to 3.3]
Statistical Analysis 7: Comparison: Everolimus 10 mg + Exemestane 25 mg vs Everolimus 10 mg; Global Satisfaction; Test type: Other; Mean Difference (Net) = -2.7, 90% CI 2-sided [-8.3 to 2.9]
Statistical Analysis 8: Comparison: Everolimus 10 mg + Exemestane 25 mg vs Capecitabine 1250 mg/m2; Global Satisfaction; Test type: Other; Mean Difference (Net) = -3.3, 90% CI 2-sided [-8.4 to 1.9]

9. Post Hoc Outcome: All Collected Deaths
Description: On treatment deaths were collected from FPFT up to 30 days after study drug discontinuation, for a maximum duration of 224 weeks (treatment duration ranged from 1.3 to 220.0 weeks).
  Deaths post treatment survival follow up were collected after the on- treatment period, up to approximately 5 years. Patients who didn't die during the on-treatment period and had not stopped study participation at the time of data cut-off (end of study) were censored.
Time Frame: up to 224 weeks (on-treatment), up to approximately 5 years (study duration)
Population: Clinical database population; all treated patients
Measure: Count of Participants; unit: Participants
Arm/Group | Everolimus 10 mg + Exemestane 25 mg | Everolimus 10 mg | Capecitabine 1250 mg/m2
Number analyzed (Participants) | 104 | 103 | 102
Participants
  On-treatment deaths | 9 | 5 | 2
  Post-treatment deaths | 62 | 55 | 57
  All deaths | 71 | 60 | 59

ADVERSE EVENTS:
Time Frame: Adverse events were collected from First Patient First Treatment (FPFT) up to 30 days after study drug discontinuation, for a maximum duration of 224 weeks (treatment duration ranged from 1.3 to 220.0 weeks).
Description: Any sign or symptom that occurs during the study treatment and 30 days post treatment follow up.
  Maximum exposure to study treatments = 201 weeks (Everolimus + Exemestane treatment group), 145 weeks (Everolimus treatment group) and 220 weeks (Capecitabine treatment group).
Arm/Group | Everolimus 10 mg + Exemestane 25 mg | Everolimus 10 mg | Capecitabine 1250 mg/m2
All-Cause Mortality (participants affected / at risk) | 9/104 | 5/103 | 2/102
Serious Adverse Events (participants affected / at risk) | 37/104 | 30/103 | 30/102
Other Adverse Events (participants affected / at risk) | 103/104 | 100/103 | 99/102
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Everolimus 10 mg + Exemestane 25 mg (N=104) | Everolimus 10 mg (N=103) | Capecitabine 1250 mg/m2 (N=102)
Anaemia (Blood and lymphatic system disorders) | 1 | 3 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Pancytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0
Cardiac arrest (Cardiac disorders) | 1 | 0 | 0
Cardiac failure (Cardiac disorders) | 1 | 0 | 0
Cardiac failure acute (Cardiac disorders) | 1 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 1 | 0
Cardio-respiratory arrest (Cardiac disorders) | 1 | 1 | 0
Pericardial effusion (Cardiac disorders) | 1 | 0 | 0
Vertigo positional (Ear and labyrinth disorders) | 1 | 1 | 0
Diplopia (Eye disorders) | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 2 | 0 | 2
Ascites (Gastrointestinal disorders) | 0 | 1 | 1
Colitis (Gastrointestinal disorders) | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 2 | 3
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 0 | 0 | 1
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 1
Gastric haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Ileus (Gastrointestinal disorders) | 1 | 0 | 0
Large intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 3 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 2 | 1
Vomiting (Gastrointestinal disorders) | 2 | 1 | 3
Death (General disorders) | 1 | 0 | 0
Drug intolerance (General disorders) | 0 | 0 | 1
Fatigue (General disorders) | 1 | 0 | 2
General physical health deterioration (General disorders) | 4 | 0 | 0
Hernia (General disorders) | 0 | 1 | 0
Multiple organ dysfunction syndrome (General disorders) | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 2 | 0 | 0
Oedema peripheral (General disorders) | 0 | 1 | 0
Performance status decreased (General disorders) | 0 | 1 | 0
Bile duct obstruction (Hepatobiliary disorders) | 0 | 1 | 0
Hepatic failure (Hepatobiliary disorders) | 2 | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 1
Bacterial pyelonephritis (Infections and infestations) | 1 | 0 | 0
Ear infection (Infections and infestations) | 1 | 0 | 0
Erysipelas (Infections and infestations) | 0 | 0 | 1
Escherichia sepsis (Infections and infestations) | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 1 | 1
Infected cyst (Infections and infestations) | 1 | 0 | 0
Infection (Infections and infestations) | 0 | 1 | 0
Lung infection (Infections and infestations) | 1 | 0 | 1
Pneumocystis jirovecii pneumonia (Infections and infestations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 8 | 4 | 2
Pyelonephritis (Infections and infestations) | 1 | 0 | 0
Sepsis (Infections and infestations) | 1 | 0 | 0
Septic shock (Infections and infestations) | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 3 | 1 | 1
Urosepsis (Infections and infestations) | 0 | 0 | 1
Fibula fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Ilium fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 0
Blood triglycerides increased (Investigations) | 1 | 0 | 0
Blood uric acid increased (Investigations) | 1 | 0 | 0
Body temperature increased (Investigations) | 1 | 0 | 0
Ejection fraction decreased (Investigations) | 0 | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 1 | 0 | 0
Platelet count decreased (Investigations) | 1 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 1 | 3
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 | 1 | 0
Failure to thrive (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 2
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Mobility decreased (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2 | 0
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 0 | 1
Hypoaesthesia (Nervous system disorders) | 1 | 0 | 0
Seizure (Nervous system disorders) | 0 | 0 | 1
Syncope (Nervous system disorders) | 2 | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 3 | 4 | 2
Nephrolithiasis (Renal and urinary disorders) | 0 | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 1
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 1
Skin toxicity (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 4
Hypotension (Vascular disorders) | 0 | 0 | 3
Hypovolaemic shock (Vascular disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Everolimus 10 mg + Exemestane 25 mg (N=104) | Everolimus 10 mg (N=103) | Capecitabine 1250 mg/m2 (N=102)
Anaemia (Blood and lymphatic system disorders) | 32 | 26 | 22
Neutropenia (Blood and lymphatic system disorders) | 4 | 4 | 14
Thrombocytopenia (Blood and lymphatic system disorders) | 4 | 7 | 3
Dry eye (Eye disorders) | 2 | 1 | 7
Lacrimation increased (Eye disorders) | 3 | 4 | 9
Abdominal pain (Gastrointestinal disorders) | 10 | 9 | 13
Abdominal pain upper (Gastrointestinal disorders) | 6 | 3 | 6
Constipation (Gastrointestinal disorders) | 14 | 15 | 18
Diarrhoea (Gastrointestinal disorders) | 36 | 34 | 55
Dry mouth (Gastrointestinal disorders) | 10 | 11 | 12
Dyspepsia (Gastrointestinal disorders) | 8 | 5 | 7
Mouth ulceration (Gastrointestinal disorders) | 15 | 13 | 1
Nausea (Gastrointestinal disorders) | 35 | 21 | 52
Stomatitis (Gastrointestinal disorders) | 51 | 45 | 24
Toothache (Gastrointestinal disorders) | 5 | 6 | 1
Vomiting (Gastrointestinal disorders) | 20 | 14 | 29
Asthenia (General disorders) | 25 | 9 | 24
Fatigue (General disorders) | 39 | 32 | 34
Non-cardiac chest pain (General disorders) | 6 | 4 | 5
Oedema peripheral (General disorders) | 30 | 22 | 16
Pyrexia (General disorders) | 18 | 12 | 9
Pneumonia (Infections and infestations) | 6 | 7 | 2
Rash pustular (Infections and infestations) | 6 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 8 | 8 | 5
Urinary tract infection (Infections and infestations) | 12 | 8 | 5
Alanine aminotransferase increased (Investigations) | 16 | 10 | 6
Aspartate aminotransferase increased (Investigations) | 16 | 14 | 9
Blood cholesterol increased (Investigations) | 6 | 9 | 1
Blood creatinine increased (Investigations) | 8 | 6 | 4
Gamma-glutamyltransferase increased (Investigations) | 15 | 16 | 2
Platelet count decreased (Investigations) | 8 | 1 | 1
Weight decreased (Investigations) | 31 | 25 | 15
Decreased appetite (Metabolism and nutrition disorders) | 35 | 32 | 27
Dehydration (Metabolism and nutrition disorders) | 9 | 5 | 5
Hypercholesterolaemia (Metabolism and nutrition disorders) | 3 | 9 | 3
Hyperglycaemia (Metabolism and nutrition disorders) | 13 | 18 | 8
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 5 | 15 | 9
Hypokalaemia (Metabolism and nutrition disorders) | 11 | 6 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 11 | 16 | 13
Back pain (Musculoskeletal and connective tissue disorders) | 20 | 8 | 12
Bone pain (Musculoskeletal and connective tissue disorders) | 9 | 4 | 7
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3 | 6 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 10 | 7 | 8
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 11 | 5 | 9
Myalgia (Musculoskeletal and connective tissue disorders) | 6 | 4 | 3
Neck pain (Musculoskeletal and connective tissue disorders) | 6 | 1 | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 14 | 13 | 16
Dizziness (Nervous system disorders) | 8 | 9 | 6
Dysgeusia (Nervous system disorders) | 17 | 20 | 14
Headache (Nervous system disorders) | 17 | 16 | 13
Neuropathy peripheral (Nervous system disorders) | 1 | 1 | 7
Paraesthesia (Nervous system disorders) | 6 | 2 | 3
Anxiety (Psychiatric disorders) | 6 | 2 | 5
Depression (Psychiatric disorders) | 8 | 5 | 5
Insomnia (Psychiatric disorders) | 10 | 8 | 11
Dysuria (Renal and urinary disorders) | 6 | 1 | 3
Breast pain (Reproductive system and breast disorders) | 6 | 1 | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 37 | 16 | 18
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 18 | 19 | 17
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 13 | 11 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 | 7 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4 | 5 | 6
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 22 | 21 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 6 | 3 | 6
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 7 | 4 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 11 | 6 | 14
Erythema (Skin and subcutaneous tissue disorders) | 6 | 4 | 3
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 3 | 3 | 62
Pruritus (Skin and subcutaneous tissue disorders) | 11 | 8 | 7
Rash (Skin and subcutaneous tissue disorders) | 22 | 23 | 12
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 | 0 | 6
Hypertension (Vascular disorders) | 15 | 8 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Statistical Analysis Plan (2017-10-27): https://cdn.clinicaltrials.gov/large-docs/44/NCT01783444/SAP_000.pdf
  • Study Protocol (2017-04-18): https://cdn.clinicaltrials.gov/large-docs/44/NCT01783444/Prot_001.pdf